CLINICAL TRIAL: NCT07228728
Title: A Randomised Controlled Trial to Investigate How Regular Skin Massage Impacts the Immune System in Early Life
Brief Title: Exploring the Cutaneous Immune Response to Skin Massage in Early Life
Acronym: CUTIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Rosetrees Trust (Other); Stoneygate Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 173023; CF-2021-2\108 (Other Grant/Funding Number: RoseTrees Trust and Stoneygate Trust)
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-10

CONDITIONS: Skin Massage
Keywords: Massage; Early life; dermatology; Immune System; Immune Response; Infant Development; Skin barrier; Microbiome; Interstitial Skin fluid
MeSH Terms: interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No application of product and no massage (No Intervention): No application of product and no massage.
- Twice-Weekly Massage with Product (Experimental): Application of product containing oil- and aqueous-based components + skin massage twice a week
  Interventions: Other: Skin Massage with Product
- Daily Massage with Product (Experimental): Application of product containing oil- and aqueous-based components + skin massage daily
  Interventions: Other: Skin Massage with Product

INTERVENTIONS:
Other: Skin Massage with Product — Application of product containing oil- and aqueous-based components to baby's skin followed by a standardized massage.
  Arms: Daily Massage with Product; Twice-Weekly Massage with Product

SUMMARY:
This project aims to study whether regular skin massage in babies induces cutaneous inflammation and whether this inflammatory response is amplified in those receiving daily (vs bi-weekly or no) skin massage over an 8 week period. Specifically, it aims to:

1. Establish if massage increases /decreases immune signals in the skin.
2. Clarify if the effects of massage are enhanced with the frequency of massage. 3.) Assess changes in skin biology as a consequence of skin massage. 4.) Determine if massage impacts skin barrier function in the early years of life.

DETAILED DESCRIPTION:
Massaging the skin is thought to be beneficial to facilitate bonding between babies and their caregivers. Evidence shows that it can help blood flow and may also positively impact the baby's immune system. However, this has not been researched in detail before. In our study, we aim to understand how the skin immune system reacts to massage. We aim to establish if regular skin massage induces cutaneous immune system changes measured through pro-inflammatory cytokines in interstitial fluid (ISF), and whether this response is amplified in those receiving daily (vs bi-weekly or no) skin massage over an 8 week period.

How skin massage influences the cutaneous immune system has not been investigated to date. The study will aim to address the following hypotheses:

1. Regular skin massage generates immune "warning" signals (such as cytokines), the precondition of the skin during healthy development, more so in those who have massaged daily (compared to no massage and bi-weekly massage).
2. Skin massage enhances skin barrier function and bacterial diversity of the skin.

The study is split into two parts. In part 1, the ISF device will be piloted in the first 9 healthy babies enrolled in the study to optimise the pressure and length of time the device is used for. Participants will be invited to attend 1 visit to the Clinical Research Facility at St Thomas' Hospital, lasting approximately 1 hour for this non-invasive collection of skin fluid and skin barrier measurements. We can offer allergy testing to house dust mite, peanut, egg and milk for your baby, if you are interested.

Part 2 is a randomised controlled trial that will investigate how regular skin massage impacts the immune system in 100 healthy baby's. Participants will be randomly allocated to 1 of 3 groups for the 8 week period:

* Group 1 (control group): No moisturiser (emollient) will be applied to your baby's skin, and they will not receive any massage.
* Group 2: You will apply a moisturiser (emollient) with oil and water-based components and massage your baby's skin twice a week.
* Group 3: You will apply a moisturiser (emollient) with oil and water-based components and massage your baby's skin daily.

Participants will be asked to attend 3 visit to the Clinical Research Facility at St Thomas' Hospital, at baseline, Week 4 and Week 8 for some non-invasive skin assessments, including skin fluid (ISF) sampling, skin barrier measurements, skin swabs, tape strips and a skin prick allergy test to house dust mite, egg, peanut and milk.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy babies born at term up to 6 months old
2. Ability of parents/guardians/caregivers to provide written informed consent for study participation
3. Willingness of parents/guardians/caregivers to comply with all study requirements.

Exclusion Criteria:

1. Parents/guardians/caregivers unable to give informed consent.
2. Personal history of inflammatory skin disease (in particular atopic dermatitis)
3. Active involvement in another interventional research study

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 109 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Detection of inflammatory cytokine markers in ISF. | 8 weeks
  The release of allergy-related and barrier-related soluble mediators such as IL-10 and TGF-β as well as other Th1/Th2 and other inflammatory cytokines.

SECONDARY OUTCOMES:
Detection of skin biology changes in ISF using genetic profiling (RNA sequencing) and proteomics. | 8 weeks
  RNA will be extracted on the ISF samples using a commercial kit. Quantification of gene expression profile will be performed with a Nanostring nCounter Analysis system. This will be used to assess panels of genes associated with allergy and inflammation. Proteomics will be conducted using mass spectrometry.
Detection of changes in barrier function | 8 weeks
  TEWL, a validated measure of skin barrier function, will be measured using a closed chamber TEWL instrument (Biox Aquaflux Model AF200) adjacent to the ISF sampling site.
To measure specific IgE to foods and aeroallergens | 8 weeks
  SPT to egg, milk, peanut and house dust mite.
To detect signals of skin microbiota e.g. bacterial diversity in addition to specific strains such as Staphylococci. | 8 weeks
  Skin microbiome swabs for microbial DNA extraction, next generation or shotgun sequencing to identify bacteria or other micro-organisms (such as viruses and fungi) will be taken. We will sample the skin flora at a 4cm2 site. The swab will be taken from the site of ISF sampling. The sample will be collected using an Isohelix® microbial DNA swabs moistened with two drops of normal saline. A (negative) control sample will be taken for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Flohr, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St. Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided